CLINICAL TRIAL: NCT05576935
Title: The Individual Response of Healthy Individuals to Mental Fatigue: a Randomized Crossover Trial Investigating the Influence of Internal Factors in the Effects of Mental Fatigue on Human Performance
Brief Title: The Individual Response of Healthy Individuals to Mental Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Bart Roelands, Professor, Vrije Universiteit Brussel
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1432022000084
Record Dates: First submitted 2022-09-07; First posted 2022-10-13 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Mental Fatigue
MeSH Terms: conditions — Mental Fatigue | interventions — Stroop Test

STUDY DESIGN:
Intervention Model Description: R randomized, single-blinded, placebo controlled, counter-balanced, cross-over design
Who Masked: Participant
Masking Description: Participants are not informed as to what condition they are subjected.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention task consists of a 60 minute Stroop task. In this task, four coloured words ("rood", "blauw", "groen" and "geel") will be presented one at a time on a computer screen. The participants will be required to indicate the colour of the word, ignoring the meaning of the word itself. If, however, the ink colour of the word is red, the button to be pressed will be the button linked to the real meaning of the word. The word presented and its ink colour will be randomly selected by a computer (100% incongruent), with all incongruent word-colour combinations being equally common. Subjects will be instructed to respond as quickly and accurately as possible. To assess performance both ACC and reaction time (RT) will be collected and averaged every block.
  Interventions: Behavioral: Stroop task
- Control (Active Comparator): In the control task subjects will have to watch a documentary of 60 min.
  Interventions: Behavioral: Documentary

INTERVENTIONS:
Behavioral: Stroop task — The task is partitioned in 4 blocks of 360 stimuli and each word will be presented on screen in 34 point font for 1000 ms with an inter-stimulus interval based on their performance on the Stroop max test. This max test will be performed during the familiarization trial, and is divided in blocks of 96 stimuli. After each block, the accuracy (ACC) will be calculated. When ACC > 85%, the difficulty of the Stroop task will be increased by decreasing the stimulus presentation time (SPT). If ACC < 85%, this block will be considered as an 'error' and the subject must redo the block without changing the SPT. The first block will have a SPT of 1500 ms. When the required ACC is achieved, the SPT will decrease in the following order: 1100, 900, 800,… to determine the individualized cognitive load. When the subject makes 3 errors in a row, or 5 errors during the whole trial, the trial will end. The SPT of the last block will be considered as the maximum capacity of that individual.
  Arms: Intervention
Behavioral: Documentary — In order to avoid under- and over-arousal, participants will have the opportunity to choose between several documentaries. The participants will also receive a list of the available documentaries (based on selections from Netflix and Disney+) after the familiarization trial so that the trial can go as smoothly as possible.
  Arms: Control

SUMMARY:
The objective of the present study is to confirm and map out the presence of interindividual differences in the effect of mental fatigue on both physical and cognitive performance, and to see if these differences are related to individual factors of the participants.

DETAILED DESCRIPTION:
Every participant will visit the lab a total of three times within a period of two weeks. In the first visit, they will undergo both a detailed screening as well as perform all intervention/control trial measures to familiarize themselves with the utilised equipment. This detailed screening entails, among other things, a maximal incremental exercise test, a cognitive test battery and multiple subjective questionnaires.

The experimental and control trial are almost identical, with the only difference being the task performed in the middel of the trial. At the beginning of the trial the EEG will be fitted to the head of the participant and baseline measures will be taken. Afterwards, participants will perform a go nogo task to assess baseline cognitive performance. Then the intervention (i.e. Stroop task) or control (i.e. documentary) task will be performed. The goal of the Stroop task is to elicit mental fatigue, while the documentary provides a meaningful comparison. Afterwards, cognitive performance will again be assessed using the go no go task, followed by a physical performance task in the form of a time trial.

The different internal factors assessed during the screening stage will be correlated to the difference in cognitive and physical performance between the intervention and control trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (No neurological, cardiovascular or musculoskeletal disorders of any kind)
* No prior knowledge of the concept of mental fatigue
* No medication
* Non-smoker

Exclusion Criteria:

* Injuries of any kind in the past 6 months
* Suffering from a chronic health condition (could be neurological, cardiovascular, internal and musculoskeletal)
* Participating in any concomitant care or research trials
* History of suffering from any mental/psychiatric disorders
* Suffering from a higher risk of burn out, indicated by a total score of ≥ 2.59 on the Burn out assessment tool (BAT)
* Suffering from high general fatigue, indicated by a score of >59 on the Multidimensional fatigue inventory (MFI)
* Suffering from depression, indicated by a score of >16 on the Beck depression inventory-II (BDI-II)
* Use of medication
* Use of caffeine and heavy efforts 24 hours prior each trial
* Suffering from colour vision deficiencies
* Not eating a standardized meal, the morning of each trial

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 142 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2024-08-23 (Actual)

PRIMARY OUTCOMES:
Physical performance | through study completion, an average of 2 years
  Participants will perform a time trial to assess physical performance. Participants will be able to start a 3 min fixed intensity warm-up. The trial itself lasts 15 min and participants are instructed to cover as much distance as possible. To keep the influence of motivation to a minimum, no encouragements or performance feedback will be given during the trial. The participants will only see the amount of time they have left on a digital chronometer. After the trial, a 2 min self-paced cooldown period will start. The evaluted outcome will be total workload performed by the participants (in kJ).
Cognitive performance: Go NoGo task: attention | through study completion, an average of 2 years
  Cognitive performance will be assessed using a task based on the go/no-go paradigm. Participants are to react to different stimuli displayed on a computer screen positioned about 1 meter from the subject, preceded by a screen with general instructions. Two different stimuli were present at the same time: a Go or NoGo stimuli, and a left or right stimuli (meaning that four combinations are possible: GoRight, GoLeft, NoGoRight and NoGoLeft). If a Go stimuli is presented, participants are instructed to react to the left or right stimuli with the corresponding arrows. However, if a NoGo stimulus is presented, participants are instructed to refrain from reacting to the either the left or right stimuli. This proposed paradigm measures attention, response inhibition and working memory. Stimuli will be presented for 500 ms, with a varying interstimulus time between 1100 and 1700 ms. Outcome for attention will be reaction time on the Go trials.
Cognitive performance: Go NoGo task: response inhibition | through study completion, an average of 2 years
  Cognitive performance will be assessed using a task based on the go/no-go paradigm. Participants are to react to different stimuli displayed on a computer screen positioned about 1 meter from the subject, preceded by a screen with general instructions. Two different stimuli were present at the same time: a Go or NoGo stimuli, and a left or right stimuli (meaning that four combinations are possible: GoRight, GoLeft, NoGoRight and NoGoLeft). If a Go stimuli is presented, participants are instructed to react to the left or right stimuli with the corresponding arrows. However, if a NoGo stimulus is presented, participants are instructed to refrain from reacting to the either the left or right stimuli. This proposed paradigm measures attention, response inhibition and working memory. Stimuli will be presented for 500 ms, with a varying interstimulus time between 1100 and 1700 ms. Outcome for response inhibition will be accuracy on the NoGo trials.

SECONDARY OUTCOMES:
Subjective Manipulation check: M-VAS | through study completion, an average of 2 years
  The M-VAS-scale (0-10cm) will be taken at multiple different time points (i.e. at the start of the trial, after the EEG baseline, after the pre cognitive performance task, after the behavioural manipulation check, during the intervention/control task, after the post behavioural manipulation check, after the post cognitive performance outcome and after the physical task). It will assess how mentally fatigued the subject is feeling (100 point VAS scale), and ranges from 'not at all' to 'completely exhausted'. The validity and reliability of a visual analogue scale to assess general fatigue was demonstrated by Lee et al., and this type of scale has been shown to be one of the most sensitive assessments of MF.
Behavioural Manipulation check: Stroop reaction time | through study completion, an average of 2 years
  Reaction time on the stroop will be assessed to determine behavioural induction of mental fatigue.
Behavioural Manipulation check: Stroop accuracy | through study completion, an average of 2 years
  Accuracy on the stroop will be assessed to determine behavioural induction of mental fatigue.
Physiological manipulation check - EEG (theta and alpha power and ERPs) | through study completion, an average of 2 years
  Electroencephalography (EEG) will be used to continuously measure brain activity by using 32 active Ag/AgCl electrodes attached on the participants' head (Acticap, Brain Products Munich, Germany), according to the "10:20 International System". The sampling rate will be set at 500 Hz (Brain Vision Recorder, Brain Products, Munich, Germany). Electrode impedance will be kept <10 kΩ throughout the recording. Baseline measurements will be taken 2 min with eyes open, 2 min with eyes closed and subjects will be seated in a sound isolated dimly lit room. Afterwards, Event-related potentials (ERP), spectral power and brain connectivity analysis will be executed. The aim of the EEG device is to measure the presence of MF during the Stroop task, and to identify possible mechanisms behind the suspected decreases in human performance.
Age | through study completion, an average of 2 years
  Age will be assessed to determine influences on mental fatigue effects
Length | through study completion, an average of 2 years
  Length will be assessed to determine influences on mental fatigue effects (using SECA 206, SECA Benelux, The Netherlands)
Weight | through study completion, an average of 2 years
  Weight will be assessed to determine influences on mental fatigue effects (using Tanita TBF 300, Tanita Europe BV, The Netherlands)
Sex | through study completion, an average of 2 years
  Sex will be assessed to determine influences on mental fatigue effects
Fat percentage | through study completion, an average of 2 years
  Fat percentage will be assessed to determine influences on mental fatigue effects (Tanita TBF 300, Tanita Europe BV, The Netherlands)
Burn out | through study completion, an average of 2 years
  General health will be assessed using the Burn out assessment tool (BAT). The questionnaire assesses 4 core domains in burn out: exhaustion, emotional impairment, cognitive impairment and mental distance Moreover, 2 additional domains that assess specific symptoms of burn out are also assessed: psychosomatic complaints and psychological distress.
Recovery need | through study completion, an average of 2 years
  Additionally, a questionnaire that determines recovery need will be added to the burn out assessment. For this part, we will use the recovery need section of the "Short Inventory to Monitor Psychosocial Hazards" questionnaire.
Physical training level (objective) | through study completion, an average of 2 years
  Objectively, a graded maximal cycle ergometer test will be performed in 18-20°C and a RH of 40%, to attain the maximal exercise ability. This ability will then be translated to a specific performance level as defined by De Pauw et al.
Physical training level (subjective) | through study completion, an average of 2 years
  Subjectively, the international physical activity questionnaire short form (IPAQ-SF) will assess the overall physical activity habits of the participant. The IPAQ-SF consists of 7 questions, assessing amount and level of intensity of physical activity in the last 7 days, and represents good reliability and validity.
Sport participation | through study completion, an average of 2 years
  a specific questionnaire will be designed with questions examining sport participation. These answers on these questions will then be employed to divide participants into a tier based system as proposed by McKay et al.
Working memory | through study completion, an average of 2 years
  Working memory will be assessed using a short n-back task. Participants will be instructed to focus on a white computer screen with a randomly generated number between 0-9. They have to press a button if the number in front of them matches the number they encountered 2 numbers earlier (2 back paradigm). Stimuli are presented for 500 ms, with an interstimulus time of 2500 ms, and a target/non target ratio of 33/67 (58). Outcomes include ACC (percentage of correct responses).
Response inhibition | through study completion, an average of 2 years
  To examine response inhibition, participants will be required to perform a sustained attention to response task (SART). Participants were presented with single digits in the centre of the screen, ranging from 0-9, and were instructed to react as fast as possible if a number was shown on screen. However, if the number that was displayed equalled 3, participants were asked to refrain from responding. To specifically measure response inhibition, the outcome of this task consisted of the percentage of correct responses to the number 3 stimulus.
Attention | through study completion, an average of 2 years
  Attention will be assessed using a psychomotor vigilance task (PVT). The task features a red triangle in the centre of a computer screen, where participants are required to react as fast as possible when a yellow count is started in the middle of this red triangle. The interstimulus time ranges between 2 and 10 sec. Mean RT is collected as outcome, and false alarms (>200 ms reaction) and misses (>900 ms) are also measured.
Genetics | through study completion, an average of 2 years
  Genes will be investigated using blood samples which will be captured in EDTA tubes and stored at -80 °C at the lab. The blood samples will be taken in between the physical assessment and the maximal incremental exercise test. One sample will then be sent to BRIGHTcore where the DNA will be extracted and analysed using exome sequencing.
Sleep quality | through study completion, an average of 2 years
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI). The PSQI's 19 self-reported items belong to one of seven subcategories: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The initial evaluation of the index found a reliability of 0.83 (good), and a test-retest reliability of 0.85 (good). Overall, the PSQI shows excellent reliability and validity for both clinical as well as non-clinical samples.
Chronotype | through study completion, an average of 2 years
  Sleep profile will be assessed using the single item chronotype scale (SIC). The SIC features six images relating to different chronotypes, and participants are required to select the picture that most closely relates to their perceived chronotype ("Which image best corresponds to your activation level during the day (i.e. in the morning, during daytime/afternoon, in the evening)?").
Trait Self control | through study completion, an average of 2 years
  Trait self-control will be assessed using brief self-control scale developed by Tangney et al.. This 13 item scale is designed to assess trait self-control and has been shown to be correlated with the total self-control scale. It supports questions such as "I am good at resisting temptation" where participants are instructed to indicate if this statement is "not at all" (1) to "very much" (5) applicable to themselves.
Trait Anxiety | through study completion, an average of 2 years
  The state-trait anxiety inventory involves two 20-item subscales describing trait and state anxiety, respectively. Only the first subscale will be used in this study. A score between 1 and 4 (from "Not at all "to "Very much so ") has to be provided on every item. The higher the score, the more severe the trait anxiety.
Mental Toughness | through study completion, an average of 2 years
  The eight item mental toughness questionnaire designed by Gucciardi et al. will be used asses MT. Participants will be asked to indicate how true each of the statements are (e.g., "I strive for continued success"), using a seven-point Likert scale (1-7) where 1 is designated as "false, 100% of the time" and 7 is designated as "true, 100% of the time".
Caffeine use | through study completion, an average of 2 years
  Will be determined using the revised caffeine consumption questionnaire (CCQ-R). This questionnaire is designed to assess the approximate self-reported consumption of caffeine during the week, with products ranging from coffee and tea to food containing caffeine and drugs, and takes about 5 min to complete. The CCQ-R is a valid way to assess caffein consumption.

OTHER OUTCOMES:
Mental workload: NASA-TLX 4 | through study completion, an average of 2 years
  Subjective workload will be measured the 4 item version of The National Aeronautics and Space Administration Task Load Index (NASA-TLX-4). The 4 item version of the NASA-TLX scale is a scale specifically designed to assess the single factor of "mental strain", as opposed to the original 6 item scale that is more a measure of general workload. Details about the original questionnaire are described by Hart and Staveland, 1988. The NASA-TLX-4 is composed of four subscales (i.e. mental demand, temporal demand, effort and frustration) and, since its task specific, will be taken after finishing the 60-min intervention/control task and after both cognitive performance outcomes. Further information on validation can be found in Hernandez et al..
Motivation: Moti-VAS | through study completion, an average of 2 years
  Motivation will be assessed using a VAS. Participants will be asked "How motivated do you feel for the upcoming task", and will be instructed to rate their answer on a 10cm line, with the statements "not at all" and "extremely motivated" at opposite ends of this line. Since motivation has often been cited as a potential mechanism behind MF, its measurement might give us a clue about the mechanisms behind possible influencing individual factors. Moreover, multiple MF studies have already used a VAS as a measuring method for motivation.
Mood: BRUMS | through study completion, an average of 2 years
  The Brunel Mood Scale (BRUMS) will be used to indicate mood, and serve as a control measure for both arousal as well as boredom . It will be assessed before and after each trial. This scale is based on the Profile of Mood States, and was validated using a multi-sample confirmatory factor analysis. It features 24 mood descriptors (divided into 6 subscales (i.e. anger, confusion, depression, fatigue, tension and vigor)), where participants have to give a value for every mood on a 5-point Likert scale (i.e. 0=not at all to 4 = extremely) responding to the question: "how do you feel right now?". It supports an adequate internal consistency and test-retest reliability. Moreover, it has been used in multiple MF studies and can accurately be used as a possible confounder variable.
Subjective physical fatigue: P-VAS | through study completion, an average of 2 years
  a P-VAS scale (0-10 cm) will be administered before, during (every 3 min) and at the end of each time trial to check the level of subjective physical fatigue of the participants. Participants will be asked to rate their general physical fatigue on a 10 cm line ranging from "not at all" to "completely exhausted". The validity and reliability of a visual analogue scale to assess general fatigue was demonstrated by Lee et al.
Sleepiness: Karolinska | through study completion, an average of 2 years
  The Karolinska Sleepiness Scale (KSS) will be conducted at the start of every trial, and before and after the intervention/control trial. This 10-point scale measures the subjective level of sleepiness and goes from 1 = 'extremely alert' to 10 = 'extremely sleepy, falls asleep all the time'. It is an often used scale in sleepiness research, Kaida et al. stated that this scale has a high validity in measuring sleepiness.
Subjective feelings of boredom: B-VAS | through study completion, an average of 2 years
  To assess the feeling of boredom the question "How boring did you find the performed task?" will be asked, the subjects will have to answer on a visual analogue scale that ranges from 'not at all' to 'completely bored'. This visual analogue scale for boredom (B-VAS) will be taken after each cognitive task, the intervention/control trial and the physical task. The validity and reliability of a general visual analogue scale has already been determined, and the B-VAS has also already been used in MF research.
Internal load | through study completion, an average of 2 years
  the internal load of the physical performance measure will be examined using the CR100 RPE scale. This scale is a valid and modified version of the original Borg RPE measure, depicting a scale of 1-100 with verbal anchors reading "nothing at all", "minimum", "extremely weak", "very weak", "weak", "moderate", "strong", "very strong", "extremely strong" and "maximal". These verbal anchors are subsequently divided into larger categories (i.e. "just noticeable", "light", "heavy", "max"). Moreover, an "absolute maximum" is also depicted, which is displayed far above the so called maximum. The CR100 scale is a reliable and valid measure of internal load in physical performance, and is hypothesized to be more sensitive to changes in internal load compared to the CR10 scale.The RPE will be examined before, after and throughout (2 min intervals) the time trial.
Glucose concentration (mmol/l) | through study completion, an average of 2 years
  Glucose concentration (mmol/l) (Bayer Contour Next USB Glucosemeter, Leverkusen, Germany) will be measured both before and after the cognitive- and physical outcome tasks. Subject's will be asked to give a 0.6-µl sample of whole blood from the left index finger top for assessment.
Heart rate | through study completion, an average of 2 years
  Heart Rate will be assessed by using the Equivital™ Life Monitor EQ-02 Physiological Status Monitor (PSM). Heart rate will be assessed during each run of the go/NoGo taks, every block of the Stroop task and the entirety of the time trial. Data will be averaged over each task and for every block of the Stroop task.
Lactate concentration (mmol/l) | through study completion, an average of 2 years
  blood lactate will be continuously measured every 3 min during the performed time trial and at the beginning and end of the trial at the right ear lobe of the participant (determined enzymatically; EKF; BIOSEN 5030, Magdeburg, Germany). It will also always be measured at the beginning and end of the physical task.

CONTACTS AND LOCATIONS:
Locations (1):
- BLITS-Brussels Labo voor Inspanning en Topsport, Etterbeek, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Yes
External users can only access the data on request and with approval from the responsible researchers, and requires a data use agreement.
  Requests will be handled directly by the responsible researchers. As mentioned, since the present study handles sensitive data, the data will not be send and saved on any external databases.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The data will become available on request as soon as the study ends. Data can be requested for at least 10 years after the end of the study.

REFERENCES:
- [Background] De Pauw K, Roelands B, Cheung SS, de Geus B, Rietjens G, Meeusen R. Guidelines to classify subject groups in sport-science research. Int J Sports Physiol Perform. 2013 Mar;8(2):111-22. doi: 10.1123/ijspp.8.2.111. PMID 23428482
- [Background] Lee KA, Hicks G, Nino-Murcia G. Validity and reliability of a scale to assess fatigue. Psychiatry Res. 1991 Mar;36(3):291-8. doi: 10.1016/0165-1781(91)90027-m. PMID 2062970
- [Background] Hernandez R, Roll SC, Jin H, Schneider S, Pyatak EA. Validation of the National Aeronautics and Space Administration Task Load Index (NASA-TLX) adapted for the whole day repeated measures context. Ergonomics. 2022 Jul;65(7):960-975. doi: 10.1080/00140139.2021.2006317. Epub 2021 Nov 22. PMID 34766872
- [Background] Kaida K, Takahashi M, Akerstedt T, Nakata A, Otsuka Y, Haratani T, Fukasawa K. Validation of the Karolinska sleepiness scale against performance and EEG variables. Clin Neurophysiol. 2006 Jul;117(7):1574-81. doi: 10.1016/j.clinph.2006.03.011. Epub 2006 May 6. PMID 16679057
- [Derived] Habay J, Arenales Arauz YL, Proost M, Schampheleer E, Lathouwers E, De Pauw K, Pattyn N, Van Cutsem J, Roelands B. Mental Fatigue Negatively Impacts Cognitive and Physical Performance Outcomes: A Large-Scale Randomized Crossover Trial. Med Sci Sports Exerc. 2026 Feb 1;58(2):225-241. doi: 10.1249/MSS.0000000000003852. Epub 2025 Sep 8. PMID 40938104